CLINICAL TRIAL: NCT00746096
Title: Phase 3, Placebo Controlled, Randomized, Double-blinded, Nonsteroidal Antiinflammatory Drug add-on Clinical Trial of Mono-phase Low Dose Oral Contraceptive Pill for Treatment of Primary Dysmenorrhea.
Brief Title: Efficacy and Safety Study of Low Dose Oral Contraceptive Pill to Treat Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IKH-01-6
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IKH-01 (Experimental): ethinyl estradiol 0.035mg and norethisterone 1mg
  Interventions: Drug: IKH-01
- Placebo (Placebo Comparator): Placebo for ethinyl estradiol 0.035mg and norethisterone 1mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IKH-01 — ethinyl estradiol 0.035mg and norethisterone 1mg
  Arms: IKH-01
Drug: Placebo — Placebo for ethinyl estradiol 0.035mg and norethisterone 1mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether combination oral contraceptive pill of norethindrone and ethinyl estradiol is effective in the treatment of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* primary dysmenorrhea

Exclusion Criteria:

* severe hepatopathy
* pregnant woman

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Terakawa, M.D.,Ph.D., Study Director — Nissay Hospital,Osaka,Japan

REFERENCES:
- [Result] Harada T, Momoeda M, Terakawa N, Taketani Y, Hoshiai H. Evaluation of a low-dose oral contraceptive pill for primary dysmenorrhea: a placebo-controlled, double-blind, randomized trial. Fertil Steril. 2011 May;95(6):1928-31. doi: 10.1016/j.fertnstert.2011.02.045. Epub 2011 Mar 21. PMID 21420678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between September 2008 and August 2009, involving 115 patients with primary dysmenorrhea at 13 center of Japan.
Groups:
- IKH-01: Patient received IKH-01 orally based on 28 days cycle that was consist of 21 days administration period and 7 days free of medication.
  The treatment was initiated on the third day of the menstrual cycle and continued to the fourth cycle.
- Placebo: Patient received placebo orally based on 28 days cycle that was consist of 21 days administration period and 7 days free of medication.
  The treatment was initiated on the third day of the menstrual cycle and continued to the fourth cycle.
Period: Overall Study
Arm/Group | IKH-01 | Placebo
Started | 58 | 57
Completed | 48 | 54
Not Completed | 10 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — No study drug treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: 58 and 57 pts were assigned to IKH-01 or placebo group, and 57 and 56 pts started study drug adminitstration. Five pts in the IKH-01 group were excluded from FAS due to no available data of efficacy but include safety set and 1 pts placebo group was exculded from FAS and safety analysis population because of no visti after the drug administration.
Groups:
- IKH-01: 0.035mg ethinyl estradiol and 1 mg norethisterone
- Total: Total of all reporting groups
Arm/Group | IKH-01 | Placebo | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (6.28) | 29.2 (7.15) | 29.1 (6.71)
Sex/Gender, Customized [Number; unit: participants]
  Female | 52 | 55 | 107
Dysmenorrhea score [Mean (Standard Deviation); unit: units on a scale] — The detail of dysmenorrhea score that was used in this study is the following. These subscales summed for a total dysmenorrhea score (minimum 0 to maximum 6). Pain score None 0 : None Mild 1 : There are some troubles for work Moderate 2 : Needing to rest in bed and/or affecting work Severe 3 : Morre than 1 day in bed and not possible to work
  Drug score (during a menstrual period) None 0 : None Mild 1 : taking analgesics for 1 days Moderate 2 : taking analgesics for 2 days Severe 3 : taking analgesics more than 3 days
  units on a scale | 3.8 (0.94) | 3.6 (0.71) | 3.7 (0.83)
VAS [Mean (Standard Deviation); unit: units on a scale] — VAS stands for Visual Analogue Scale of pain. The scale was rated as a graphic rating scale. as a 100mm baseline from 0:No pain to 100:Worst possible pain.
  units on a scale | 57.2 (18.00) | 60.0 (16.82) | 58.6 (17.32)

OUTCOME MEASURES:

1. Primary Outcome: Patient Response to Treatment for Primary Dysmenorrhea, as Evaluated by Difference of Total Dysmenorrhea Score (Baseline/Pretreatment-End of Treatment)
Description: The detail of dysmenorrhea score that was used in this study is the following. These subscales summed for a total dysmenorrhea score (minimum 0 to maximum 6). Pain score None 0 : None Mild 1 : There are some troubles for work Moderate 2 : Needing to rest in bed and/or affecting work Severe 3 : Morre than 1 day in bed and not possible to work
  Drug score (during a menstrual period) None 0 : None Mild 1 : taking analgesics for 1 days Moderate 2 : taking analgesics for 2 days Severe 3 : taking analgesics more than 3 days
Time Frame: 16weeks
Population: Five patients in the IKH-01 group were excluded from efficacy analysis due to no available data for 3 patients and 2-4 administration days for 2 patients.
  One patient in the placebo group was also excluded from efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo for 0.035mg ethinyl estradiol and 1 mg norethisterone
Arm/Group | IKH-01 | Placebo
Number analyzed (Participants) | 52 | 55
units on a scale
  Baseline (0W) | 3.8 (0.94) | 3.6 (0.71)
  End of Treatment (16W) | 1.2 (1.26) | 2.2 (1.43)

2. Secondary Outcome: Difference in the VAS of Primary Dysmenorrhea (Baseline/Pretreatment-dnd of Treatment)
Description: VAS stands for Visual Analogue Scale of pain. The scale was rated as a graphic rating scale. as a 100mm baseline from 0:No pain to 100:Worst possible pain.
Time Frame: 16weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IKH-01 | Placebo
Number analyzed (Participants) | 52 | 55
units on a scale
  Baseline (0W) | 57.2 (21.1) | 60.0 (16.82)
  End of Treatment (16W) | 21.2 (21.05) | 39.2 (23.10)

ADVERSE EVENTS:
Time Frame: From study administration to 6 cycles of menstruation, an average of 6 months
Arm/Group | IKH-01 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/55
Other Adverse Events (participants affected / at risk) | 52/57 | 40/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IKH-01 (N=57) | Placebo (N=55)
Nausea (Gastrointestinal disorders) | 8 (9) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 4 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (40) | 15 (21)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Blood triglyceride increased (Investigations) | 5 (6) | 2 (2)
Protein urine prsent (Investigations) | 4 (4) | 2 (2)
Blood fibrinogen increased (Investigations) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 6 (8)
Metrorrhagia (Reproductive system and breast disorders) | 37 (66) | 8 (21)
Oligomenorrhoea (Reproductive system and breast disorders) | 8 (12) | 8 (11)
Hypomenorrhoea (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 3 (5) | 2 (2)
Polymenorrhoea (Reproductive system and breast disorders) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.